CLINICAL TRIAL: NCT03573479
Title: Early Rehabilitation in Critically Ill Children - The PICU Lliber8 Study
Brief Title: Early Rehabilitation in Critically Ill Children - The PICU Liber8 Study
Acronym: PICULiber8
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Karen Choong, Professor, McMaster University
Other Study IDs: PICULiber8/180409
Record Dates: First submitted 2018-05-30; First posted 2018-06-29 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Delirium; Withdrawal Syndrome; Hospital Acquired Condition; Critical Illness Myopathy; Critical Illness
Keywords: rehabilitation; critical care; child health; quality improvement
MeSH Terms: conditions — Delirium; Substance Withdrawal Syndrome; Iatrogenic Disease; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation cohort: This is the pre-implementation phase where a baseline documentation will take place about usual clinical practice, perceptions and attitudes of PICU staff and clinicians
- PICU Liber8 bundle: After the implementation of the bundle (the PICU Liber8 components) same measurements will be captured and analyzed comparatively.
  Interventions: Other: PICU Liber8 Bundle

INTERVENTIONS:
Other: PICU Liber8 Bundle — Bundle of elements for quality improvement
  Other Names: implementation of strategy
  Groups: PICU Liber8 bundle

SUMMARY:
This is a pilot quality improvement implementation study that will measure the impact of a rehabilitation bundle implementation on the outcomes of interest. Advancements in the care provided in Pediatric Intensive Care Units (PICUs) have led to fewer deaths in children. These improvements are unfortunately countered by the emergence of side effects of critical illness, known as PICU-acquired complications (PACs). Delirium, muscle weakness, drug dependency and withdrawal are increasingly common. PACs occur because children are often over-sedated and experience long periods of immobilization. PACs delay recovery, increase disability and worsen long-term function and quality-of-life. Although they are preventable, PACs are very common and frequently overlooked by clinicians. This study aims to "liberate"children from critical illness and improve their recovery and functioning after discharge, through an innovative rehabilitation bundle of 8 complementary steps (PICU Liber8) to reduce sedation, allow children to awaken and breathe comfortably, encourage early mobilization, and engage families in their child's care.

DETAILED DESCRIPTION:
This is a pilot quality improvement implementation study that will measure the impact of a rehabilitation bundle.

The objectives are:

1. Primary - Implementation Objectives: to determine the feasibility and resources required to implement PICU Liber8 in 2 PICUs, evaluate strategies for successful bundle adoption. Co-Primary - Process Objectives: to determine the impact of PICU Liber8 on the process of care.
2. Secondary Efficacy: impact on PACs and patient reported outcomes The methods consist of a PICU Liber8 Bundle Implementation Plan (Pronovost's 4 E's Framework), and measurement of the impact of Implementation through Orchestrated Testing (OT).

For successful adoption of the PICU Liber8 bundle, the following are necessary:

1. A context appropriate implementation framework.
2. An implementation team leader.
3. Inter-professional team engagement (i.e. RN, RT, MD, pharmacy, allied health and family).
4. Ability to customize PICU Liber8 to the needs of each site. We will use the Pronovost's implementation framework, which has been shown to facilitate successful bundle adoption and improve the quality of patient care in adult and pediatric ICUs.17-19 This framework has 4 phases: Engage, Educate, Execute and Evaluate.

ELIGIBILITY:
Inclusion criteria: All children admitted to the Pediatric Intensive Care Unit with a minimum of 48h stay in the PICU and more than one organ dysfunction.

Exclusion criteria: as this is an assessment of a quality improvement strategy there are no criteria for excluding participants.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted to the PICU for the QI intervention. For patient follow-up we will conduct for patients at risk (see eligibility criteria)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Completion rate of daily goals (compliance) | 18 months
  The total number and percentage of daily goals completed from a pre-established daily goals checklist that assess compliance with the bundle. This is considered part of the feasibility outcomes group.
Performance of the bundle assessed with qualitative (i.e., narrative) description and comparison between groups. | 18 months
  Evaluation of performance as narrative description and comparison between periods of study, about the impact of the bundle on the process of quality of care. This also is part of the feasibility outcomes group.
Perceptions about barriers and facilitators for implementation of the bundle | 18 months
  Qualitative (i.e., narrative) assessment, description, and comparison of the perceptions from key stakeholders (i.e., family members, patients, clinicians, administrative personnel, nurse team, etc.) between groups about perceived barriers and facilitators for the adequate bundle's implementation. This belongs to the acceptability outcome.

SECONDARY OUTCOMES:
Economic analysis | 18 months
  Direct cost (in Canadian dollars) before and after the implementation of the bundle that measures activity-based costs associated with the implementation. Incremental costs of PICU associated complications will be added to this evaluation.
Incidence of morbidities | 18 months
  Measured as the composite incidence (number of new cases) of either delirium, iatrogenic withdrawal, pressure ulcers, or PICU acquired weakness.
Length of stay | 1 month
  Measured as total days in PICU and hospital, and hospital-free days at 30 days post PICU discharge.
Ventilator-free days at 30 days | 1 month
  This is a clinically important outcome, measured as days using mechanical ventilation and days without it.
30-day mortality | 18 months
  Measured as the total number of deaths (due to any cause) during the PICU and/or hospital stay.
Functionality | 18 months
  Using the Pediatric Evaluation and Disability Inventory-Computer Adaptive Test (PEDI-CAT), which measures abilities in three functional domains: Daily Activities, Mobility, and Social/Cognitive. The PEDI-CAT's Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks. A final score per several domains is calculated that ranges from 0 to 100.
Health related quality of life | 18 months
  Using the Peds-QL, which includes four Scales (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning) that are grouped together on the actual questionnaire. The tool creates a final score from 0 to 100 (higher scores indicates better).
Parental stress | 18 months
  Using the Pediatric Inventory for Parents, a 42 item score across 4 domains. Higher scores indicate greater frequency and difficulty.
Risk measurement of psychological sequelae. | 18 months
  The risk of psychological sequelae will be measured with the Children's Critical Illness Impact Scale (CCIIS) for children >6 years of age, consisting of 23 items that result on the final scale (where higher scores are worse).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MD, MSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Sciences, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be collected from both participating sites and analyzed at the coordinating centre at McMaster.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one month of completing the study.
Access Criteria: A Data Access Agreement has been completed and signed among participating centres. Further data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Choong K, Koo KK, Clark H, Chu R, Thabane L, Burns KE, Cook DJ, Herridge MS, Meade MO. Early mobilization in critically ill children: a survey of Canadian practice. Crit Care Med. 2013 Jul;41(7):1745-53. doi: 10.1097/CCM.0b013e318287f592. PMID 23507722
- [Background] Cameron S, Ball I, Cepinskas G, Choong K, Doherty TJ, Ellis CG, Martin CM, Mele TS, Sharpe M, Shoemaker JK, Fraser DD. Early mobilization in the critical care unit: A review of adult and pediatric literature. J Crit Care. 2015 Aug;30(4):664-72. doi: 10.1016/j.jcrc.2015.03.032. Epub 2015 Apr 8. PMID 25987293
- [Background] Choong K, Foster G, Fraser DD, Hutchison JS, Joffe AR, Jouvet PA, Menon K, Pullenayegum E, Ward RE; Canadian Critical Care Trials Group. Acute rehabilitation practices in critically ill children: a multicenter study. Pediatr Crit Care Med. 2014 Jul;15(6):e270-9. doi: 10.1097/PCC.0000000000000160. PMID 24777303
- [Background] Wieczorek B, Ascenzi J, Kim Y, Lenker H, Potter C, Shata NJ, Mitchell L, Haut C, Berkowitz I, Pidcock F, Hoch J, Malamed C, Kravitz T, Kudchadkar SR. PICU Up!: Impact of a Quality Improvement Intervention to Promote Early Mobilization in Critically Ill Children. Pediatr Crit Care Med. 2016 Dec;17(12):e559-e566. doi: 10.1097/PCC.0000000000000983. PMID 27759596
- [Background] Choong K, Fraser D, Al-Harbi S, Borham A, Cameron J, Cameron S, Cheng J, Clark H, Doherty T, Fayed N, Gorter JW, Herridge M, Khetani M, Menon K, Seabrook J, Simpson R, Thabane L. Functional Recovery in Critically Ill Children, the "WeeCover" Multicenter Study. Pediatr Crit Care Med. 2018 Feb;19(2):145-154. doi: 10.1097/PCC.0000000000001421. PMID 29394221